CLINICAL TRIAL: NCT00457184
Title: Thrombophilia and Migraine, Are They Related? - A Clinical Study
Brief Title: Thrombophilia and Migraine, Are They Related?
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 1700802.EMC
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2004-01

CONDITIONS: Migraine; Thrombosis; Thrombophilia
Keywords: Migraine; Thrombosis; Thrombophilia
MeSH Terms: conditions — Migraine Disorders; Thrombosis; Thrombophilia | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood tests

SUMMARY:
Migraine was described as related to stroke in adults and children as well. Complete thrombophilic status was not study in large groups of pediatric patients. The purpose of our study is to assess the prethrombotic profile among children and teenagers diagnosed as suffering from migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as suffering from migraine according to the Neurologic criteria.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2004-01; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit, Ha'Emek Medical Center; Miriam Kutai, MD, Principal Investigator — Pediatric Neurology Unit - Ha'Emek Medical Center
Locations (1):
- Pediatric Hematology Unit - HaEmek Medical Center, Afula, Israel